CLINICAL TRIAL: NCT05657275
Title: Impact on the Use of Antibiotics of a Multimodal Algorithm for the Diagnosis and Management of Acute Community-acquired Pneumonia in the Emergency Room
Acronym: PROMCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP221018
Record Dates: First submitted 2022-12-10; First posted 2022-12-20 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Community-acquired Pneumonia
Keywords: CRP dosage; multiplex PCR; chest scan without injection
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: Chronological series in alternating periods, that is to say alternations of periods of more or less short duration, with and without intervention corresponding to a repetition of before/after studies will be carried
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention period (Experimental): Patient management will be guided by a multimodal algorithm integrating the performance of biological and iconographic examinations
  Interventions: Diagnostic Test: CRP dosage; Diagnostic Test: multiplex PCR; Diagnostic Test: chest scan without injection
- Control period (No Intervention): Patient management will be done according to the usual practices of centers and emergency physicians

INTERVENTIONS:
Diagnostic Test: CRP dosage — multimodal algorithm
  Arms: Intervention period
Diagnostic Test: multiplex PCR — multimodal algorithm
  Arms: Intervention period
Diagnostic Test: chest scan without injection — multimodal algorithm
  Arms: Intervention period

SUMMARY:
Reducing antibiotics prescription is still to date, the main goal in low respiratory tract infections (LRTI).

Several studies have shown conflicting results on the impact of multiplex PCR as a point of care tool. Our experience has highlighted an impact on single room assignments during the winter season but not yet on antibiotics prescriptions. This project aims to evaluate a new multimodal algorithm including multiplex PCR at the point of care to reduce antibiotics prescription and therefore has the ability to have a positive impact on antibiotics resistance phenomenon.

DETAILED DESCRIPTION:
Acute community-acquired pneumonia (CAP) is the leading infectious cause of infectious death worldwide and the third leading cause of death from all causes. They are also very frequent reasons for visit to the emergency room, especially during winter season. Although respiratory viruses are responsible for approximately 30 to 50% of CAP, antibiotics' prescription remain very high. This prescription is at the origin of the phenomenon of antibiotic resistance, which continues to increase throughout the world. In the meantime, the biological testing of this clinical picture is increasingly evolving since a decade, and this evolution has been even accelerated with the emergence of COVID-19. With regard to the increasing availability of respiratory viruses testing, we need more studies allowing to better use these results to spare antibiotics when useless.

Several avenues of study have been investigated to improve the diagnosis of bacterial CAP and thus reduce unnecessary antibiotic therapy: differentiating viral CAP from bacterial CAP using multiplex PCR and/or inflammation biomarkers, localizing the infection lung parenchyma using chest CT.

The various studies carried out on the impact of the use of multiplex PCR in the emergency department (ED) led to discordant conclusions. The study carried out within Bichat Claude-Bernard Hospital only shows an interest for single room assignment in patients infected with pathogens such as influenza, RSV and Metapneumovirus. Multiplex PCR delocalized to the ED does not seem to be a sufficient measure to reduce the prescription of antibiotics in patients suspected of CAP admitted from the emergency room. One study carried during the COVID-19 pandemic highlighted that multiplex PCR, used as a point of care, induced improvements in patient flow and infection control measures.

C Reactive Protein (CRP) is a well-known inflammation biomarker. Previous studies estimate that CRP has better performance than procalcitonin in the diagnosis of pneumonia with thresholds often described at 50 mg.L-1 and revised upwards in older patients. The National Institute for Health and Care Excellence (NICE) has endorsed the use of point-of-care CRP to diagnose CAP and reduce inappropriate antibiotic use. This recent meta-analysis suggests that CRP is a better marker than PCT for the diagnosis of pneumonia. Indeed, a CRP >20 mg/L, >50 mg/L or >100 mg/L has a positive LR+ likelihood ratio of 2.08, 3.68, and 5.79, respectively, and a negative LR- likelihood ratio of 0.32, 0.36, and 0.48, while PCT >0.25 µg/L or >0.50 µg/L has an LR+ of 5.43 and 8.25, respectively, and an LR- of 0.62 and 0.76.

In addition, the place of imaging in reducing the prescription of antibiotics in CAP is still very little studied; nevertheless, CT without injection has proven to be of great help in the diagnosis of COVID-19 and remains the gold standard (reference examination) for effectively diagnosing CAP.

The current recommendations of the French society of infectious diseases do not clearly mention the use of multiplex PCR. CRP is included as a biomarker of inflammation in favor of bacterial infection when it is high. The CT scan is mentioned in cases where the diagnosis of CAP is difficult without defining the criteria for this difficult diagnosis. The College of Pneumology Teachers updated in 2020 places multiplex PCR as an essential diagnostic tool in the management of CAP. Finally, the latest American recommendations (2018) mention the performance of a multiplex PCR as indicated in any patient admitted to hospital with symptoms of influenza-like illness. As a result, the practices of hospitals are very heterogeneous in the diagnosis of CAP, we therefore propose to develop a multimodal algorithm combining multiplex PCR, CRP and chest CT scan in the diagnosis of CAP in patients requiring hospitalization, starting as soon as possible during winter.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years or older
* Presence of at least one respiratory sign among the following: dyspnea, cough, expectoration, auscultatory abnormalities, chest pain;
* Presence of at least one general sign among the following: fever (T>38°C), hypothermia (T<35°C), myalgia, headache, asthenia;
* Oxygen-requiring patient defined by a saturation <95% or presenting a risk area among:

  * Age > 65 years old
  * Alcoholic and/or tobacco intoxication
  * Congestive heart failure
  * Cerebrovascular disease (stroke or transient ischemic attack)
  * Chronic kidney disease (excluding dialysis)
  * Chronic liver disease
  * Unbalanced diabetes mellitus
  * Progressive neoplastic disease
  * Immunodepression (systemic corticosteroid therapy or immunosuppressive treatment within 6 months, splenectomy, chemotherapy within 6 months, HIV at the AIDS stage, cachexia, etc.)
  * Homozygous sickle cell disease
  * Bacterial pneumonia
  * Hospitalization during the year
  * Institutional life

Non-inclusion Criteria:

* Patient unable to consent: coma or acute respiratory distress requiring orotracheal intubation
* Patient with chronic renal failure on dialysis
* Patient with a history of chronic obstructive pulmonary disease
* Lung transplant patient
* Patient being treated with antibiotics at the time of the emergency room consultation
* Patient simultaneously participating in an interventional study protocol (assessing the duration of antibiotic therapy)
* Pregnant or breastfeeding woman
* Patient refusal to participate
* Patient deprived of freedom or under a legal protective measure
* Patient under guardianship or curatorship or with cognitive impairment
* Non-affiliation to a social security regimen or CMU

Exclusion Criteria:

• RT-PCR positive for SARS-CoV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Total duration (in days) of pulmonary-targeted antibiotic therapy | day 30

SECONDARY OUTCOMES:
Total duration of hospitalization (in days) | day 30
Proportion of patients who died within 30 days | day 30
Proportion of patients rehospitalized within 30 days | day 30
Proportion of patients hospitalized in a single room | day 30
Proportion of patients with initiation of pulmonary-targeted antibiotic treatment in the emergency department | day 1
Proportion of patients with discontinuation of pulmonary-targeted antibiotic treatment in the emergency department | day 3
Proportion of patients with initiation or discontinuation of pulmonary-targeted antibiotic treatment in medical wards or ICU. | day 30
Proportion of patients with initiation of antiviral treatment | day 30

CONTACTS AND LOCATIONS:
Overall Officials: Donia BOUZID, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - CHU Nîmes, Nîmes
  - Bichat hospital, Paris

IPD SHARING:
Plan to Share IPD: No